CLINICAL TRIAL: NCT06720883
Title: Robotically Assisted Surgery For Perihilar Cholangiocarcinoma: A Prospective Study
Acronym: ROBOCHOL
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Prof. Umberto Cillo, Azienda Ospedaliera di Padova
Other Study IDs: AOP3105
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cholangiocarcinoma Cancer; Perihilar Cholangiocarcinoma
Keywords: cholangiocarcinoma; robot; robotic; perihilar; cca; phc
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma; Congenital contractural arachnodactyly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — liver samples, lymphnodes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients affected by pCCA requiring curative intent robotic surgery with biliary reconstruction: All patients affected by pCCA candidate for curative intent robotic liver resection with biliary reconstruction will be enrolled in the study after the work up for surgery. Preoperative, intraoperative and postoperative data will be collected. The DaVinci® robotic platform available at the Padova University hospital will be utilised primarily. We will include patients with age≥18 years, with histologically proven pCCA or highly presumed bile duct malignancy with difficulties to obtain histological evidence with negative Immunoglobulin G4 (IgG4 sample). We will not include patients with distant metastases, previous radiotherapy, vascular encasement, ASA score>4, synchronous malignancy in other organs or indication for palliative surgery
  Interventions: Procedure: Major hepatectomy

INTERVENTIONS:
Procedure: Major hepatectomy — All patients will undergo robotic major hepatectomy with S1 resection, hilar lymphadenectomy and biliary reconstruction

SUMMARY:
Cholangiocarcinoma (CCA) represents the most common biliary tract malignancy, and the second most common primary hepatic malignancy, accounting for 15% to 20% of primary liver tumours.

Perihilar cholangiocarcinoma (pCCA) involves the biliary confluence with or without involvement of the right and left hepatic ducts. Complete resection with negative histologic margins is the only chance of cure and the most robust predictor of long-term survival for patients affected by any type of locally advanced CCA. However, the proximity of perihilar tumors to vital structures makes curative excision technically difficult.

Minimally invasive approaches are progressively spreading in liver surgery units worldwide. Significant advantages of minimally invasive liver resections, if compared to open one, have been diffusely shown, such as shorter hospital stay and possibility of complex reconstructive procedures similar to those performed in open surgery. Robot-assisted liver surgery represents a natural consequence of such a minimally invasive evolution.

This is a monocentric, single arm, observational, prospective study that aims at analyzing the outcomes of robotic major liver resection and biliary recontruction for perihilar cholangiocarcinoma.

Among study outcomes, the primary outcome is evaluation of morbidity; secondary outcomes includes conversion rate, margin status, biliary fistula, liver failure, disease specific survival, overall Survival

Data related to patient condition (laboratory tests, etc.), surgery performed, and post-surgical course will be collected.

The protocol for this study has been developed in accordance with the European Union Good Clinical Practice guidelines and the Declaration of Helsinki, and it has been approved by the Territorial Ethics Committee of the East-Central Veneto Area (CETAEV).

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) represents the most common biliary tract malignancy, and the second most common primary hepatic malignancy, accounting for 15% to 20% of primary liver tumours. The incidence of bile duct cancers is increasing worldwide, currently accounting for 3% of all gastrointestinal cancers (1).

According to the anatomical location it is classified as follows: intrahepatic (iCCA), perihilar (pCCA) and distal (dCCA) subtypes. Approximately 50% of CCA are perihilar, 40% are extrahepatic and only 10% or less are intrahepatic (2). Each type of cholangiocarcinoma is characterised by differences in the tumour biology and management, each has a separate American Joint Committee on Cancer (AJCC) staging system (2).

Perihilar cholangiocarcinoma (pCCA), also called Klatskin tumour, involves the biliary confluence with or without involvement of the right and left hepatic ducts (3, 4, 5). It is a challenging disease to manage in the preoperatory setting and during surgery. Painless jaundice is the main symptom at presentation. It often arises rapidly and it is present in 90% of pCCA. Fatigue, anorexia, weight loss and non-specific abdominal pain are other common symptoms.

Complete resection with negative histologic margins is the only chance of cure and the most robust predictor of long-term survival for patients affected by any type of locally advanced CCA. However, the proximity of perihilar tumors to vital structures, such as the hepatic artery, portal vein, and hepatic parenchyma, makes curative excision technically difficult.

Median survival for patients who cannot undergo surgery is 12 months. Patients who receive radical surgical resection have a 5-year survival up to 40% (6, 7).

Radical surgical resection of pCCA usually requires a hemi-hepatectomy, often extended. For this reason, the preoperative assessment of the future liver remnant volume (FLR) is a critical step in the surgical plan. Traditionally, a "safe" liver resection requires a FLR of at least 25% in a perfectly healthy liver. When the organ is compromised by steatosis, chronic cholestasis, cirrhosis or chemotherapy this rate has to increase up to 40% (8, 9). Regional lymphnode metastases are not considered an absolute contraindication to resection, although N+ disease is an independent prognostic factor for worse outcome. Nevertheless, complete lymphadenectomy of the hepatoduodenal ligament is considered an essential step of the surgical procedure.

Liver and bile duct resection for pCCA are technically complex procedures: the specimen resection with negative margins requires careful dissection of major vascular structures such as portal vein and hepatic arteries. Once completed the resection the biliary tract must be reconstructed, usually with a Jejunal loop. This step of the procedure is particularly complex and requires high levels of skills and detail, thus, so far, has widely limited the use of laparoscopic surgery to complete the surgical procedure.

As previously in other fields of surgery, minimally invasive approaches are progressively spreading in liver surgery units worldwide. Significant advantages of minimally invasive liver resections, if compared to open one, have been diffusely shown. In particular, lower morbidity and shorter hospital stays have been demonstrated in many numerically relevant series. Interestingly enough, greater advantages compared to open surgery have been shown in cases of "laparoscopically difficult" liver resections as right or left hepatectomy. Robot-assisted liver surgery represents a natural consequence of such a minimally invasive evolution. Potential advantages of Robot assisted approach are "intuitive". In particular, in liver surgery the relationship between instrument angle of incidence and plans of action occurs in spatially complex and extremely variable scenarios. More than in other surgical settings, such an articulated spatial interaction needs flexible and harmonic movements warranted in robot assisted interventions.

Recent evidence confirms Robot assisted hepatectomies are associated with less postoperative pain and shorter hospital stay if compared to open liver resections. At the same time, both minor and major Robot assisted hepatectomies showed similar oncologic performance, morbidity and mortality profile than open liver resections (10, 11). The key advantage of robotic assistance is to allow complex reconstructive procedures similar to those performed in open surgery (12). The relevant developments already achieved in the field of pancreatic surgery (13) are paradigmatic with relevant future perspectives. Indeed, the Whipple reconstruction phase is now performed in many leading robotic assisted HPB centres. It is easy to predict that in hepatobiliary surgery as well the next steps of development will include major vasculo-biliary reconstructions.

AIM OF THE STUDY The aim of the study is investigating the potential advantage of Robotic major liver surgery with biliary reconstruction for pCCA utilising a robotic platform, such as the DaVinci® robotic platform, currently available at the Padova teaching hospital and in use for the HPB service.

OUTCOMES Primary Outcomes Morbidity: Defined as major and minor complication rate according to Dindo-Clavien classification (14) and Comprehensive Complication Index (CCI), including ninety-days mortality

Secondary Outcomes

* Conversion rate
* Margin status (R0 Vs R1)
* Biliary Fistula: As defined by International Study Group of Liver Surgery (15)
* Liver failure: As defined by International Study Group of Liver Surgery (16)
* Disease specific survival
* Overall Survival (1-3-5 years)

STUDY POPULATION AND METHODS This is a prospective observational study. All patients affected by pCCA that will undergo curative intent surgery that requires biliary reconstruction will be enrolled in the study after the work up for surgery. Preoperative, intraoperative and postoperative data will be collected. The DaVinci® robotic platform available at the Padova University hospital will be utilised primarily. In case of future acquisition of newer or different robotic platforms, those will be utilised as well for the study. The postoperative outcome, morbidity, mortality, pathologic margins, number of lymph nodes collected, and long-term oncologic outcome will be reviewed and compared with the historical cohort of the HPB service of Padova University that includes more than 150 cases completed after 2004.

INCLUSION CRITERIA Age≥18 years Histologically proven pCCA Highly presumed bile duct malignancy with difficulties to obtain histological evidence with negative Immunoglobulin G4 (IgG4 sample) Preoperative staging work up performed by abdomen enhanced CT scan. The subject understands the nature of this trial and is willing to comply. Ability to provide written informed consent. Patients treated with curative intent in accordance to international guidelines

EXCLUSION CRITERIA Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs.

Previous radiotherapy Vascular encasement Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score>4.

Synchronous malignancy in other organs. Palliative surgery

Pathologic Evaluation All surgical specimens will be submitted for histopathological evaluation by adopting a standardised protocol where only dedicated pathologists with expertise in gastro-intestinal pathology will assess the specimens. To adequately determine residual disease status, five resection planes (common bile duct, proximal bile duct, hepatic artery, portal vein, and liver parenchyma) and one periductal dissection plane will be obtained from each surgical specimen. Histological reports will include the following clinicopathological parameters: tumor's size and differentiation grade, vascular, perineural and intraductal invasion, resection/dissection planes status, tumor growth pattern (mass forming, periductal infiltrating, intraductal, and mixed type), lymph node status and coexisting pathology (inflammation, fibrosis, steatosis, sclerosing cholangitis etc.). The annular resection margins (common bile duct, proximal bile duct, hepatic artery, and portal vein) will be recorded as positive or negative, since their slices are generally 1 to 3 mm thick and a "negative" annular plane ensures a margin of > 1 mm. For non-annular planes (periductal and liver parenchyma), margins will be assessed as positive if cancer is up to 1 mm along the dissection plane in the hepatoduodenal ligament or on the liver transection plane. The presence of severe dysplasia or carcinoma in situ at the surgical margin will be classified as a negative margin. The final pathological staging will be generated according to the revised American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) TNM staging system 8th edition (17).

Statistical analysis Values for categorical variables will be expressed as totals and percentages whereas for continuous variables they will be expressed as medians and ranges or interquartile ranges. Statistical analyses will be performed using the Pearson's chi-squared test or Fisher's test for categorical variables such as Liver failure biliary leakage hemorrhage and other complications and the Kruskal-Wallis rank sum test for continuous variables, such as length of hospital stay, intensive care length of stay etc.

The length of follow-up will be calculated from the date of surgery to the date of patient death (overall survival-OS) or the latest follow-up. The durations of follow-up and survival will be expressed as medians (interquartile ranges). Survival and recurrence curves will be calculated using the Kaplan-Meier technique and compared with the log-rank test. A p value < 0.05 will be considered to indicate statistical significance, variables with a p value < 0.1 were considered of marginal statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Histologically proven pCCA or highly presumed bile duct malignancy with difficulties to obtain histological evidence with negative Immunoglobulin G4 (IgG4 sample)
* Preoperative staging work up performed by abdomen enhanced CT scan.
* The subject understands the nature of this trial and is willing to comply.
* Ability to provide written informed consent.
* Patients treated with curative intent in accordance to international guidelines

Exclusion Criteria:

* Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs.
* Previous radiotherapy
* Vascular encasement
* Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score>4.
* Synchronous malignancy in other organs.
* Palliative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by pCCA that will undergo curative intent robotic major liver resection that requires biliary reconstruction will be enrolled in the study after the work up for surgery. Preoperative, intraoperative and postoperative data will be collected. The DaVinci® robotic platform available at the Padova University hospital will be utilised primarily.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2027-07-07 (Estimated); Study Completion 2031-07-07 (Estimated)

PRIMARY OUTCOMES:
Morbidity | From surgery to 90-days after surgery
  Defined as major and minor complication rate according to Dindo-Clavien classification and Comprehensive Complication Index (CCI), including ninety-days mortality

SECONDARY OUTCOMES:
Conversion rate | Day of surgery
  Conversion is defined as the transition from robot-assisted surgery to open surgery and is measured by calculating the percentage ratio between the number of conversions and the total number of procedures performed.
Margins status | Day of surgery
  All surgical specimens will be submitted for histopathological evaluation by adopting a standardised protocol where only dedicated pathologists with expertise in gastro-intestinal pathology will assess the specimens. To adequately determine residual disease status, five resection planes (common bile duct, proximal bile duct, hepatic artery, portal vein, and liver parenchyma) and one periductal dissection plane will be obtained from each surgical specimen. The annular resection margins (common bile duct, proximal bile duct, hepatic artery, and portal vein) will be recorded as positive or negative, since their slices are generally 1 to 3 mm thick and a "negative" annular plane ensures a margin of > 1 mm. For non-annular planes (periductal and liver parenchyma), margins will be assessed as positive if cancer is up to 1 mm along the dissection plane in the hepatoduodenal ligament or on the liver transection plane.
Biliary fistula | From surgery to 90 days after surgery
  As defined by International Study Group of Liver Surgery, drain/serum bilirubin ratio > 3 at day 3
Liver failure | From surgery to 90 days after surgery
  As defined by International Study Group of Liver Surgery, the deterioration (increase in INR and bilirubin levels) in the synthesis, excretion, and detoxification functions of the liver after liver surgery (day 5 or later)
Diseases specific survival | From surgery to 5 years after surgery
  This outcome is defined as the proportion of patients who remain alive for a specific period after robotic surgery for pCCA , without dying from cholangiocarcinoma or complications of the oncological disease
Overall Survival | From surgery to 5 years after surgery
  Overall Survival is defined as the length of time from robotic surgery for pCCA until death from any cause, and it will be evaluated at 1 year from surgery, 3 years from surgery, 5 years from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD can be provided by the principal investigator upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting information will be available from 07/07/2027 till 07/07/2031